CLINICAL TRIAL: NCT03148106
Title: Optimizing Peripheral Stimulation Parameters to Modulate the Sensorimotor Cortex for Post-stroke Motor Recovery.
Brief Title: Hand Rehabilitation Study for Stroke Patients
Acronym: DOSES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-12346; R01MH111871 (NIH)
Record Dates: First submitted 2017-03-08; First posted 2017-05-10 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Upper Extremity Paresis; Disability Physical; Chronic Stroke; Motor Disorders
MeSH Terms: conditions — Paresis; Motor Disorders | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Somatosensory Electrical Stimulation (Experimental)
  Interventions: Device: Somatosensory Electrical Stimulation

INTERVENTIONS:
Device: Somatosensory Electrical Stimulation — The investigators will put adhesive electrodes on the affected arm and connect it to a device that will deliver a gentle electrical stimulation to the hand and arm. The stimulation will last for different amounts of time, depending on the stimulation condition. This can be 30 minutes twice a day (1 hour apart), 1 hour continuously, 2 hours continuously, or 3 hours continuously. The stimulation conditions will also vary in stimulation strength. It is normal that some people may feel a tingling sensation, while others may feel nothing.
  Other Names: transcutaneous electrical nerve stimulation

SUMMARY:
The purpose of this study is to find out what are the best settings for applying electrical nerve stimulation over the skin for the short-term improvement of hand dysfunction after a stroke. The ultimate goal is to some day design an effective long-term training program to help someone recovery their ability to use their hands and function independently at home and in society. In order to know how to apply electrical nerve stimulation to produce a good long-term effect on hand dysfunction, the investigators first need to know how to make it work best in the short-term, and improve our understanding of for whom it works and how it works. The investigators will use a commercially available transcutaneous electrical nerve stimulation (TENS) unit to gently apply electrical nerve stimulation over the skin of the affected arm. This is a portable, safe and easy to use device designed for patients to operate in their homes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years, has residual hand motor dysfunction caused by a single ischemic and/or hemorrhagic stroke greater than 6 months prior to enrollment.

Exclusion Criteria:

* Pregnant; uncontrolled medical problems including but not limited to severe cardiovascular and cardiopulmonary disease; active cancer; significant hand joint deformity or other diagnosis with major effect on hand function besides stroke; severe alcohol or drug abuse within the past year; untreated or inadequately treated major depression; spasticity score >3 on the MAS; lack of finger range of motion of at least 10 degrees; severe aphasia or other communicative, behavioral or cognitive impairment that significantly interferes with the participant's ability to comply with the protocol or provide informed consent. In addition, patients will be excluded if they have a pacemaker.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Finger Fractionation | Baseline and immediately post-stimulation
  Ability to fractionate movement can be assessed by asking the patient to move one segment in isolation and keep other, adjacent segments still.

SECONDARY OUTCOMES:
Change in Modified Ashworth Scale | Baseline and immediately post-stimulation
  standard instrument
Change in Arm Research Action Test | Baseline and immediately post-stimulation
  standard instrument

CONTACTS AND LOCATIONS:
Overall Officials: Karunesh Ganguly, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No